CLINICAL TRIAL: NCT02624713
Title: Development of Eating Disorders Symptoms Among Children Who Took Part in Family-based Obesity Treatment and Among Their Siblings
Brief Title: Development of Eating Disorders Symptoms Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Hai College (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Principal Investigator, suzan berman, principal investigator, Tel Hai College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: telhaicollege
Record Dates: First submitted 2015-11-18; First posted 2015-12-08 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Eating Disorders Symptoms
Keywords: eating disorder; childhood obesity; family based treatment
MeSH Terms: conditions — Feeding and Eating Disorders; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This research is an open clinical study with two branches: a retrospective follow up and a prospective follow up
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retrospective Random Controlled Research (Other): In the controlled retrospective follow up, (not random) 44 families participated with their 81 children and siblings. The intervention group included 18 families who participated in the "Maccabi Active" program (obesity treatment) in the years 2012-2013 in the northern district, with their 24 children (18 overweight children and 6 siblings). The control group included 26 families with their 57 children (27 children who had been overweight or obese in the years 2012-2013 when they were 8-14 years old and their 30 siblings). These families did not take part in a family based treatment for their overweight child. The parameters were measured at one set point time. All participants from both the control and research groups were evaluated at the follow-up and the data collected at follow-up is being reported collectively for the Retrospective Controlled Research branch.
  Interventions: Behavioral: obesity treatment
- The Prospective study (Other): The Prospective study had only an intervention group (obesity treatment). Forty-two families took part in this study, with 78 children: 48 overweight children and 30 siblings . The parameters were measured in three different times. Before the program (time 1), at the end of the program (after 6 months - time 2) and 8 months after completing the program (time 3).
  Interventions: Behavioral: obesity treatment

INTERVENTIONS:
Behavioral: obesity treatment — 1. Parents' education groups for nutrition and healthy behavior with a dietician and a social worker every 2 weeks for5 months, for a total of 10 meetings. This part of the intervention aimed at providing parents with effective tools for modification of lifestyle and the family environment.
  2. Children's individual therapy consisted of 6 individual meetings with a family physician, a physical therapist specializing in children's physical activity, and a dietician. This part of the intervention aimed at modifying nutrition and lifestyle; the physical therapist can help children incorporate physical activity into their routine.
  3. Physical activity groups for the children, with individual physical fitness monitoring. twice a week for 6 months. .
  Other Names: family based obesity treatment

SUMMARY:
Randomized Clinical Trial, the research will be composed of two parts in order to examine the research question: a combination of controlled randomized retrospective research and prospective cohort research

Prospective Cohort Research:

The research groups - families coming for treatment in "Active Maccabi" clinics in the Northern Region, Israel. Approximately 30 families.

Retrospective Random Controlled Research

1. The research group - families that have completed an intervention program of "Active Maccabi" Northern Region, Israel,within the past two to three years. The families will be requested to attend a follow-up meeting of all family members in which they will answer questionnaires. Approximately 66 families.
2. The control groups - families who did not participate in the program who have a child between the age 7-14 who has suffered from obesity/weight (over the past 2-3 years), in correlation with the child in the intervention group. Approximately 66 families.

Hypotheses of the research:

1. Status of the weight of the child being treated and of his siblings will be higher than that at the end of the program.
2. Indication of the obesogenic environment of families participating in the program will be lower in comparison with families not participating in the program.
3. The rate of eating disorder symptoms among children who participated in the program will be lower in comparison with those of the obese/overweight child in families who were not the program.
4. The rate of eating disorder symptoms among siblings who participated in the program will be lower than that of siblings in families not in the program.

DETAILED DESCRIPTION:
Duration of the Research -Prospective Cohort Research: 6 months of intervention. 8 months follow-up.

Research Instruments

1. Anthropometric measurements of all children in the family (height, weight and BMI). BMI per centile examinations according to age.
2. An acquaintance questionnaire and demographic details - to be answered by parents
3. A FEAQ_R questionnaire to be answered by the parents (only in the prospective research group). The questionnaire will examine the obesogenic burden in the family. A column will be added for each sibling of relevant age. The questionnaire will be valid in English and Hebrew. The psychometric characteristics of the questionnaire: Alpha cronbach - validity 0.84; Reliability 0.78 Trt
4. Eat-26 (cheat) questionnaire to be answered by the children and their siblings. The questionnaire will examine the risk of developing an eating disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Families who participated in "Active Maccabi
2. Families who signed a consent form
3. Families who attended 80% of the sessions

exclusion criteria:

1. Families who don't fill in questionnaires at all stages of the research
2. Families in which the parents refuse to sign a consent form
3. Families in the control group who receive treatment in more than three sessions by a dietician in the community

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2015-11; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moria Golan, PROFESSOR, Principal Investigator — Tel Hai College

REFERENCES:
- [Background] Endevelt R, Elkayam O, Cohen R, Peled R, Tal-Pony L, Michaelis Grunwald R, Valinsky L, Porath A, Heymann AD. An intensive family intervention clinic for reducing childhood obesity. J Am Board Fam Med. 2014 May-Jun;27(3):321-8. doi: 10.3122/jabfm.2014.03.130243. PMID 24808110
- [Background] Epstein LH, Paluch RA, Raynor HA. Sex differences in obese children and siblings in family-based obesity treatment. Obes Res. 2001 Dec;9(12):746-53. doi: 10.1038/oby.2001.103. PMID 11743058
- [Background] Golan M, Crow S. Targeting parents exclusively in the treatment of childhood obesity: long-term results. Obes Res. 2004 Feb;12(2):357-61. doi: 10.1038/oby.2004.45. PMID 14981230
- [Background] Golan M, Fainaru M, Weizman A. Role of behaviour modification in the treatment of childhood obesity with the parents as the exclusive agents of change. Int J Obes Relat Metab Disord. 1998 Dec;22(12):1217-24. doi: 10.1038/sj.ijo.0800749. PMID 9877257
- [Background] Golan M, Weizman A. Reliability and validity of the Family Eating and Activity Habits Questionnaire. Eur J Clin Nutr. 1998 Oct;52(10):771-7. doi: 10.1038/sj.ejcn.1600647. PMID 9805227
- [Background] Maloney MJ, McGuire JB, Daniels SR. Reliability testing of a children's version of the Eating Attitude Test. J Am Acad Child Adolesc Psychiatry. 1988 Sep;27(5):541-3. doi: 10.1097/00004583-198809000-00004. No abstract available. PMID 3182615

RESULTS

PARTICIPANT FLOW:
Groups:
- Prospective Study: The Prospective study had only an intervention group. The intervention group included families who participated in the "Maccabi Active" program in 2015 in the northern district. The parameters were measured in three different times. Before the program (time 1), at the end of the program (after 6 months - time 2) and 8 months after completing the program (time 3). Anthropometric measurements were taken and a Cheat 26 questionnaire was given to each child in the families. The parents filled personal details and a questionnaire for mapping the family eating habits (FEAHQ-33).
- Retrospective Controlled Research: Retrospective Controlled Research The research group - families that have completed an intervention program of "Active Maccabi" Northern Region, Israel,within the past two to three years. The families will be requested to attend a follow-up meeting of all family members in which they will answer questionnaires..
  The control groups - families who did not participate in the program who have a child between the age 7-14 who has suffered from obesity/weight (over the past 2-3 years), in correlation with the child in the intervention group.
  All participants from both the control and research groups were evaluated at the follow-up and the data collected at follow-up is being reported collectively for the Retrospective Controlled Research branch.
Period: Overall Study
Arm/Group | Prospective Study | Retrospective Controlled Research
Started | 78 | 81
Completed | 64 | 81
Not Completed | 14 | 0
Not completed — Lost to Follow-up | 14 | 0

BASELINE CHARACTERISTICS:
Population: Obesity treatment: 78 children Retrospective Random Controlled Research Group: 81 children
Groups:
- Prospective Study: obesity treatment: 1.Parents' education groups for nutrition and healthy behavior with a dietitian and a social worker every 2 weeks for 5 months, for a total of 10 meetings. This part of the intervention aimed at providing parents with effective tools for modification of lifestyle and the family environment. 2. Children's individual therapy consisted of 6 individual meetings with a family physician, a physical therapist specializing in children.
- Retrospective Random Controlled Research: Retrospective Random Controlled Research
  1. The research group - families that have completed an intervention program of "Active Maccabi" ,within the past two to three years. The families will be requested to attend a follow-up meeting of all family members in which they will answer questionnaires. Approximately 66 families.
  2. The control groups - families who did not participate in the program who have a child between the age 7-14 who has suffered from obesity/weight (over the past 2-3 years), .
- Total: Total of all reporting groups
Arm/Group | Prospective Study | Retrospective Random Controlled Research | Total
Number analyzed (Participants) | 78 | 81 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 78 | 81 | 159
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 39 | 88
  Male | 29 | 42 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With >20 on the 26 Children Eating Attitudes Test
Description: Children Eating Attitudes Test- 26 items. The Children Eating Attitudes has been validated for children and adolescents. The items are rated on a 6-point scale: (1) never, (2) rarely, (3) sometimes, (4) often, (5) usually, and (6) always. Scores range from 0 (minimum) to 78 (maximum). Scores above 20 indicates a high level of concern about dieting, body weight, or problematic eating behaviors. Higher scores (above 20) are considered a worse outcome.
Time Frame: Before the program (time 1), at the end of the program (after 6 months - time 2) and 8 months after completing the program (after a total of 14 months from baseline, time 3)"
Measure: Count of Participants; unit: Participants
Groups:
- Obesity Treatment: Retrospective Random Controlled Research
  1. The research group - families that have completed an intervention program of "Active Maccabi" ,within the past two to three years. The families will be requested to attend a follow-up meeting of all family members in which they will answer questionnaires. Approximately 66 families.
  2. The control groups - families who did not participate in the program who have a child between the age 7-14 who has suffered from obesity/weight (over the past 2-3 years), .
  obesity treatment: 1.Parents' education groups for nutrition and healthy behavior with a dietician and a social worker every 2 weeks for5 months, for a total of 10 meetings. This part of the intervention aimed at providing parents with effective tools for modification of lifestyle and the family environment. 2. Children's individual therapy consisted of 6 individual meetings with a family physician, a physical therapist specializing in children's physi
- Prospective Research: Forty-two families took part in this study, with 78 children: 48 overweight children and 30 siblings. The parameters were measured in three different times. Before the program (time 1), at the end of the program (after 6 months - time 2) and 8 months after completing the program (time 3). Anthropometric measurements were taken and the Eat 26 questionnaire was given to each child in the families. The parents filled personal details and answered questions regarding the family eating habits.
Arm/Group | Obesity Treatment | Prospective Research
Number analyzed (Participants) | 81 | 78
Participants | 26 | 4

2. Primary Outcome: Family Eating and Activity Habits Questionnaire 32
Description: Family Eating and Activity Habits questionnaire (FEAHQ-32) filled out by the participating parents (only in the prospective research group). The FEAHQ is a 32-item self-report instrument designed to assess the eating and activity habits of family members as well as obesogenic factors in the overall home environment (stimulus and behaviour patterns) related to weight. The higher the score, the greater the obsogenic load in a family so its a worse outcome. The lower the score, the less obsogenic load in the family so its a better outcome. There is no minimum or maximum score as reported by Golan & Weizman, 1998 (See reference 5). The score varies from family to family according to the number of persons.The goal is to get a lower score relative to the initial score. The FEAHQ-32 has been validated in English and Hebrew.
  This measure was only used to assess the Prospective Research group, as also mentioned under research instruments in the detailed study description.
Time Frame: as for outcome 1
Population: 42 Parents answered the questionnaire before and after the program, and follow up.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Prospective Research: Forty-two families (one parent in each family) took part in this study, with 78 children: 48 overweight children and 30 siblings. The parameters were measured in three different times. Before the program (time 1), at the end of the program (after 6 months - time 2) and 8 months after completing the program (time 3). Anthropometric measurements were taken and the Eat 26 questionnaire was given to each child in the families. The parents filled personal details and answered questions regarding the family eating habits.
Arm/Group | Prospective Research
Number analyzed (Participants) | 42
score on a scale
  Difference between time 2 and time 1 | -16.2 (4.9)
  Difference between time 3 and time 2 | -23.2 (5.7)

ADVERSE EVENTS:
Groups:
- Prospective Study: Obesity research
  1. Parents' education groups for nutrition and healthy behavior with a dietitian and a social worker every 2 weeks for 5 months, for a total of 10 meetings. This part of the intervention aimed at providing parents with effective tools for modification of lifestyle and the family environment.
  2. Children's individual therapy consisted of 6 individual meetings with a family physician, a physical therapist specializing in children's physi
- Retrospective Random Controlled Research: Retrospective Random Controlled Research
  1. The research group - families that have completed an intervention program of "Active Maccabi" ,within the past two to three years. The families will be requested to attend a follow-up meeting of all family members in which they will answer questionnaires. Approximately 66 families.
  2. The control groups - families who did not participate in the program who have a child between the age 7-14 who has suffered from obesity/weight (over the past 2-3 years)
Arm/Group | Prospective Study | Retrospective Random Controlled Research
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/81
Other Adverse Events (participants affected / at risk) | 0/78 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No